CLINICAL TRIAL: NCT04468932
Title: Cerebellar Transcranial Magnetic Stimulation for Motor Control in Progressive Supranuclear Palsy
Brief Title: Transcranial Magnetic Stimulation in Progressive Supranuclear Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center of Neuromodulation for Rehabilitation (Other); Collins Medical Trust (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Department of Health and Human Services (U.S. Federal Agency); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Marian L Dale, MD, Associate Professor of Neurology, School of Medicine; Director, OHSU CurePSP Center of Care, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY0020341; KL2TR002370 (NIH); P2CHD086844 (NIH); K23NS121402 (NIH)
Record Dates: First submitted 2020-07-07; First posted 2020-07-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Palsy Supranuclear; Supranuclear Palsy, Progressive
Keywords: repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The investigators will use a single-blind crossover design with a 4 week TMS washout period. The subjects will serve as their own controls, thus limiting confounding variables such as medication or cognitive effect.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The subjects will be blinded to the order of intervention, but the PI will not be blinded in order to perform the TMS intervention. The outcome evaluators will be blinded to the intervention, however.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS first (Experimental): After completing their baseline assessment, participants randomized to this arm will initially take part in a 2-week TMS intervention. After the midpoint assessment and subsequent a 1-month washout, these participants will then complete a 2-week sham TMS period prior to their final assessment.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Sham treatment first (Experimental): After completing their baseline assessment, participants randomized to this arm will initially take part in a 2-week sham TMS period. After the midpoint assessment and subsequent a 1-month washout, these participants will then complete a 2-week TMS intervention prior to their final assessment.
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — Aim 1: To determine the clinical effects of rTMS targeting the cerebellum on postural instability in PSP. The hypothesis to be tested is that TMS augmentation of cerebellar inhibition will improve cerebellum-dependent balance symptoms of PSP for a period of time sufficient to improve rehabilitation outcomes. The investigators will measure a battery of objective posturography metrics and other measures of motor control, including sway and center of pressure changes to backward tilt and forward translation.
  Aim 2: We will use functional near infrared spectroscopy (fNIRS) to examine changes in motor and premotor cortical activity after cerebellar rTMS. The hypothesis to be tested is that premotor and motor cortical activity will decrease after cerebellar rTMS compared to sham TMS, reflecting improved cerebellar inhibition of the motor cortex after the intervention.

SUMMARY:
The objective of this proposal is to investigate the effect of non-invasive repetitive cerebellar transcranial magnetic stimulation (rTMS) on motor control in progressive supranuclear (PSP). The central hypothesis is that augmenting cerebellar inhibition via cerebellar rTMS will decrease postural instability in patients with PSP. We will use functional near infrared spectroscopy (fNIRS) to examine changes in motor and premotor cortical activity after cerebellar rTMS.

ELIGIBILITY:
Inclusion Criteria:

* probable or possible PSP by the revised MDS PSP Criteria (Hoglinger 2017)
* age 40-85 at time of screening
* ability to understand and cooperate with simple instructions in English
* ability to read at 6th grade reading level in English
* ability to stand unassisted for at least 30 seconds and to be able walk independently with a walker
* ability to refrain from new physical and speech therapy programs for the duration of the study
* ability to remain on stable doses of any cholinergic, dopaminergic, serotonergic sedative or NMDA receptor antagonists for the duration of the study
* females of child-bearing age must perform a urine pregnancy test and be on reliable birth control during the course of the study

Exclusion Criteria:

* other significant neurological or vestibular disorders
* presence of electrically, magnetically or mechanically activated implants or history of injurious metal exposure in eyes, head, or body

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
objective posturography | assessed on 4 days during the 8 week study period
  The primary endpoint is center of pressure shifts with tilt and with translation, and body sway in quiet stance.

SECONDARY OUTCOMES:
fNIRS | assessed on 4 days during the 8 week study period
  functional near infrared spectroscopy of premotor and motor areas during balance testing
speech analysis | assessed on 4 days during the 8 week study period
  speech sample assessment conducted by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Marian L Dale, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No